CLINICAL TRIAL: NCT05562050
Title: Characteristics of the Anosmic Olfactory Mucosa
Status: Active, not recruiting | Type: Observational
Sponsor: Nicolai Nielsen (Other)
Responsible Party: Sponsor-Investigator, Nicolai Nielsen, Medical doctor, Regional Hospital West Jutland
Organization: Regional Hospital West Jutland (Other)
Other Study IDs: 1-10-72-106-22
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Anosmia; COVID-19; Head Injury
MeSH Terms: conditions — Anosmia; COVID-19; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control
- COVID-19 related anosmia
- Head-trauma related anosmia

SUMMARY:
The present study aims to describe the structural tissue and cell characteristics of the olfactory mucosa in patients with persistent anosmia (≥2 years) due to COVID-19 or head-trauma, in comparison to healthy individuals with intact olfactory function. In order to avoid possible age-related degenerative changes in the neuro-epithelium, both patients and controls are between 25 and 35 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent to vouch for their own study participation.
* Informed and written consent for participation in this study.
* Study group 1 (Post-COVID anosmia)

  1. Diagnosed with persistent anosmia for approximately two years concurring with positive SARS-CoV-2 PCR-test between 2019 and 2020.
  2. Sniffin'sticks test with a threshold-discrimination-identification-score(TDI)≤16
  3. Between 25 and 35 years of age.

Study group 2 (Post-trauma anosmia)

1. Diagnosed with persistent anosmia for approximately two years concurring with head trauma.
2. Sniffin'sticks test with a threshold-discrimination-identification-score(TDI)≤16
3. Between 25 and 35 years of age.

Study group 3 (Controls):

1. Between 25 and 35 years of age.
2. Undergoing reposition of a nasal fracture in general anaesthesia

Exclusion Criteria:

* <25 years of age.
* >35 years of age.
* Chronic rhinosinusitis with/without polyps.
* Nasal cancer.
* Presence of viral or bacterial rhinosinusitis.
* Uncontrolled allergic rhinosinusitis.
* Coagulation deficiencies, e.g. haemophilia.
* Use of anticoagulants.
* Not able to undergo general anaesthesia.
* Pregnancy.
* Any use of nasal detumescence drugs ≤2 weeks before biopsy.
* Any use of nasal steroids ≤3 months before biopsy.
* Use of nasal inhaled recreational drugs ≤3 month before biopsy.
* Participants not able to communicate in Danish or English.
* Major Depression Inventory (MDI) score ≥27 [49, 50]
* Mini Mental State Examination (MMSE) score ≤ 26 [51]
* Study group 1 (Post-COVID anosmia)

  1. Anosmia for less than two years or more than two and a half years.
  2. No positive SARS-CoV-2 PCR-test concurring with olfactory dysfunction.
  3. History of olfactory dysfunction before COVID-19 infection.
* Study group 2 (Post-trauma anosmia)

  1. Anosmia for less than two years or more than approximately two-three years.
  2. Anosmia without concurring with head trauma
  3. History of prior olfactory dysfunction before head trauma.
* Study group 3 (Controls) 1. Known olfactory dysfunction.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: recruited from the clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Histological evaluation | 2023-2024
  density
Immunohistochemical evaluation | 2023-2024
  density

CONTACTS AND LOCATIONS:
Overall Officials: Therese Ovesen, DMSc, Principal Investigator — Gødstrup Hospital
Locations (1):
- ENT department, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Yes